CLINICAL TRIAL: NCT01128686
Title: A Retrospective Cohort Study to Evaluate the Rate of Good Responses to Lamivudine (LAM) Treatment in naïve Chronic Hepatitis B (CHB) Patients With Certain Pre-treatment Characteristics
Brief Title: Lamivudine(LAM) Good Responder Study
Acronym: LAMGR
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113973
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B, Chronic
Keywords: retrospective; naïve Chronic Hepatitis B (CHB) patients; cohort study; lamivudine
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CHB patients who started LAM as an initial antiviral treatment: CHB patients who started LAM as an initial antiviral treatment at least 5 years prior to this investigation
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This study is retrospective chart review

SUMMARY:
This is to evaluate the proportion of subjects who show good responses to LAM treatment in Korea.

DETAILED DESCRIPTION:
This is to evaluate the proportion of subjects who show good responses to LAM treatment such as HBV DNA negativity, HBV DNA less than 4 log, no resistant mutation, HBeAg seroconversion and normalization of ALT in naïve CHB patients with certain pre-treatment characteristics, i.e. HBV DNA less than 9log copies per ml and ALT more than 2 times ULN in HBeAg positive subjects, HBV DNA less than 7log copies per ml and elevated ALT in HBeAg negative subjects.

ELIGIBILITY:
Inclusion Criteria:

1. CHB or liver cirrhosis due to Hepatitis B virus who had started LAM between Jan 1, 2003 and Dec 31, 2004 and maintained LAM at least 6 months
2. HBsAg positive at least for 6 months at the beginning of observation
3. HBV DNA positive before LAM administration
4. Subjects with certain pre-treatment laboratory findings as follows; HBV DNA less than 9log copies per ml and ALT more than 2 times ULN in HBeAg positive patients, HBV DNA less than 7log copies per ml and elevated ALT in HBeAg negative patients

Exclusion Criteria:

1. Documented co-infection with HCV, HIV at the beginning of LAM treatment
2. Decompensated liver cirrhosis at the beginning of LAM treatment
3. HCC at the beginning of LAM treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CHB patients who started LAM as an initial antiviral treatment at least 5 years prior to this investigation in General Hospital
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects showing HBV DNA negativity at 5 years of LAM treatment | 5years

SECONDARY OUTCOMES:
Proportion of subjects showing HBV DNA negativity during first 4 years of LAM treatment | 4 years
Proportion of subjects showing HBV DNA less than 4 log copies per ml during 5 years of LAM treatment | 5 years
Cumulative proportion of subjects showing HBeAg seroconversion during 5 years of LAM treatment | 5 years
Cumulative proportion of subjects showing HBeAg loss during 5 years of LAM treatment | 5 years
Proportion of subjects showing ALT normalization during 5 years of LAM treatment | 5 years
Cumulative proportion of subjects showing resistant mutation during 5 years of LAM treatment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Kangwon-do, South Korea